CLINICAL TRIAL: NCT01927640
Title: Study of Dexmedetomidine for the Reversal of Cocaine's Effects on Myocardial Perfusion
Brief Title: Dexmedetomidine for Reversal of Cocaine's Effects on the Heart
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Lincy Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro19549
Record Dates: First submitted 2013-08-19; First posted 2013-08-22 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2018-04

CONDITIONS: Chest Pain; Acute Coronary Syndrome
Keywords: Cocaine; Dexmedetomidine; Myocardial Contrast Echocardiography
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine and intranasal cocaine (Experimental): Intranasal cocaine administration (2 mg/kg) then Dexmedetomidine (0.3-0.6 mcg/kg) infusion
  Interventions: Drug: Dexmedetomidine; Drug: Intranasal cocaine
- Normal saline and intranasal cocaine (Placebo Comparator): Intranasal cocaine administration (2 mg/kg) then Saline (over 10 minutes I.V. infusion)
  Interventions: Drug: Normal Saline; Drug: Intranasal cocaine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine (0.3-0.6 mcg/kg) infusion.
  Other Names: Precedex
  Arms: Dexmedetomidine and intranasal cocaine
Drug: Normal Saline — Normal saline infusion (10 cc)
  Arms: Normal saline and intranasal cocaine
Drug: Intranasal cocaine — Intranasal cocaine (2 mg/kg)

SUMMARY:
This study will use myocardial contrast echocardiography performed during a continuous intravenous infusion of Definity microbubbles (Perflutren lipid microbubbles) to determine if dexmedetomidine (an intravenous central sympatholytic drug) can reverse all the cardiovascular effects of low-dose intranasal cocaine-including vasoconstriction in the coronary microcirculation-both in cocaine-naïve and non-treatment seeking cocaine-addicted subjects.

DETAILED DESCRIPTION:
Each subject will be participating in three study visits: Screening Visit, Visit 1: a low-dose dobutamine visit and Visit 2: a low-dose cocaine visit. At the dobutamine visit, the subject will only receive low-dose dobutamine, which will be used as an internal inotropic/vasodilator control for cocaine. At the cocaine visit, the subject will receive low-dose intranasal cocaine followed by either the active study drug (dexmedetomidine) or an inactive placebo (saline). Both cocaine and dobutamine will increase myocardial contractility and oxygen demand, thereby stimulating metabolic vasodilation. If, as predicted, cocaine also causes α-adrenergic agonist in the coronary microcirculation, then myocardial blood flow should increase less with cocaine then with dobutamine for a given level of myocardial oxygen demand. We will study if dexmedetomidine, a central sympatholytic, can normalize this cocaine effect. We previously have used dobutamine as a comparator for cocaine in our research. At both visits, myocardial contrast echocardiography will be used to measure regional myocardial perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects ages of 18-65 years without any history of substance abuse (other than tobacco), including narcotics, abuse of prescription painkillers, cocaine or any other recreational drug

Exclusion Criteria:

* Known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts or detected by screening echocardiogram performed prior to I.V. infusion of Definity microbubbles
* Hypersensitivity or prior reactions to Definity microbubbles
* Pregnant or nursing women
* Any evidence of cardiopulmonary disease by history or physical examination, including subjects who are taking any cardiovascular medications of any sort
* History of hypertension or BP at time of consent > 140/90 mm Hg
* Any history of substance abuse (other than tobacco), including narcotics, prescription painkillers, cocaine or any other recreational drug (any person that says they have EVER tried these drugs will be excluded from this study)
* Subjects reporting alcohol intake of more than 2 drinks/day
* Severe psychiatric illness (e.g., schizophrenia, suicidal depression) in addition to drug dependence, which may signify a high risk of addiction
* Diabetes mellitus or any other systemic illness
* Individuals with a history of pseudocholinesterase deficiency
* Hypersensitivity to dexmedetomidine or lorazepam
* The presence of alcohol by breathalyzer
* Subjects who have poor echocardiography images will be screen failed.
* Persons with mechanically, magnetically, or electrically activated implants, such as cardiac pacemakers, neurostimulators, and infusion pumps (MRI only).
* Persons with ferromagnetic implants and ferromagnetic foreign bodies, such as intracranial, aneurysm clips, shrapnel and intraocular metal chips as these could become dislodged (MRI only).
* Persons unable to tolerate MRI imaging secondary to an inability to lie supine or severe claustrophobia (MRI only).
* Persons whose renal function test does not meet CSMC standard of care MRI contrast protocol requirements (GFR <45ml/min).
* Persons with allergy to animal dander or animal-instigated asthma
* Persons with a history of kidney or liver disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-01-15 (Actual); Study Completion 2014-01-15 (Actual)

PRIMARY OUTCOMES:
Myocardial Perfusion | Baseline and Immediately after acute administration of study drug (Day 1)
  Myocardial perfusion will be measured by myocardial contrast echocardiography after dexmedetomidine administration and compared to baseline. There will be no repeat dosing of dexmedetomidine. No longer term outcomes are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai, Los Angeles, California, United States

REFERENCES:
- [Background] Kontak AC, Victor RG, Vongpatanasin W. Dexmedetomidine as a novel countermeasure for cocaine-induced central sympathoexcitation in cocaine-addicted humans. Hypertension. 2013 Feb;61(2):388-94. doi: 10.1161/HYPERTENSIONAHA.112.203554. Epub 2013 Jan 2. PMID 23283356
- [Background] Menon DV, Wang Z, Fadel PJ, Arbique D, Leonard D, Li JL, Victor RG, Vongpatanasin W. Central sympatholysis as a novel countermeasure for cocaine-induced sympathetic activation and vasoconstriction in humans. J Am Coll Cardiol. 2007 Aug 14;50(7):626-33. doi: 10.1016/j.jacc.2007.03.060. Epub 2007 Jul 30. PMID 17692748
- [Background] Tuncel M, Wang Z, Arbique D, Fadel PJ, Victor RG, Vongpatanasin W. Mechanism of the blood pressure--raising effect of cocaine in humans. Circulation. 2002 Mar 5;105(9):1054-9. doi: 10.1161/hc0902.104714. PMID 11877354
- [Background] Crandall CG, Vongpatanasin W, Victor RG. Mechanism of cocaine-induced hyperthermia in humans. Ann Intern Med. 2002 Jun 4;136(11):785-91. doi: 10.7326/0003-4819-136-11-200206040-00006. PMID 12044126
- [Background] Vongpatanasin W, Mansour Y, Chavoshan B, Arbique D, Victor RG. Cocaine stimulates the human cardiovascular system via a central mechanism of action. Circulation. 1999 Aug 3;100(5):497-502. doi: 10.1161/01.cir.100.5.497. PMID 10430763
- [Background] Jacobsen TN, Grayburn PA, Snyder RW 2nd, Hansen J, Chavoshan B, Landau C, Lange RA, Hillis LD, Victor RG. Effects of intranasal cocaine on sympathetic nerve discharge in humans. J Clin Invest. 1997 Feb 15;99(4):628-34. doi: 10.1172/JCI119205. PMID 9045864